CLINICAL TRIAL: NCT03936777
Title: An Open-Label Extension Trial to Assess the Long-Term Safety of ZX008 (Fenfluramine Hydrochloride) Oral Solution as an Adjunctive Therapy for Seizures in Patients With Rare Seizure Disorders Such as Epileptic Encephalopathies Including Dravet Syndrome and Lennox-Gastaut Syndrome
Brief Title: A Study to Investigate the Long-Term Safety of ZX008 (Fenfluramine Hydrochloride) Oral Solution in Children and Adults With Epileptic Encephalopathy Including Dravet Syndrome and Lennox-Gastaut Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zogenix, Inc. (Industry)
Collaborators: Zogenix International Limited, Inc., a subsidiary of Zogenix, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZX008-1900; 2019-001331-31 (EudraCT Number); U1111-1309-4338 (Other: World Health Organization (WHO)); 2024-515680-61 (Registry Identifier: EU Clinical Trials)
Record Dates: First submitted 2019-04-12; First posted 2019-05-03 (Actual); Results first posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Dravet Syndrome; Lennox Gastaut Syndrome; Epileptic Encephalopathy
MeSH Terms: conditions — Epilepsies, Myoclonic; Lennox Gastaut Syndrome | interventions — Fenfluramine

STUDY DESIGN:
Intervention Model Description: Single Group Assisgnment
Masking Description: None (open label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ZX008 (Fenfluramine Hydrochloride) (Experimental): ZX008 is supplied as an open-label oral solution.Doses will include up to 0.8 mg/kg/day divided into 2 daily doses, up to a maximum of 30 mg/day (subjects taking concomitant STP will receive up to 0.5 mg/kg/day, up to a maximum of 20 mg/day) in a concentration of 2.5 mg/mL.
  Interventions: Drug: ZX008 (Fenfluramine Hydrochloride)

INTERVENTIONS:
Drug: ZX008 (Fenfluramine Hydrochloride) — Fenfluramine hydrochloride provided in a concentration of 2.5 mg/mL.

SUMMARY:
This is an international, multicenter, open-label, long-term safety study of ZX008 in subjects with Dravet syndrome, Lennox-Gastaut syndrome or epileptic encephalopathy

DETAILED DESCRIPTION:
This is an international, multicenter, open-label, long-term safety study of ZX008 in patients with epileptic encephalopathy, including Dravet syndrome or Lennox-Gastaut syndrome. Subjects eligible for participation are those with Dravet syndrome who are currently enrolled in Study ZX008-1503, or those with Lennox-Gastaut syndrome who have successfully completed Study ZX008-1601-Part 2, and are candidates for continued treatment with ZX008 for an extended period of time, or those with Dravet syndrome, Lennox-Gastaut syndrome, or another epileptic encephalopathy who have completed participation in another Zogenix-sponsored study and have been invited to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Male or nonpregnant, nonlactating female
* Satisfactory completion of a core study
* Has a rare seizure disorder, such as epileptic encephalopathy and has successfully completed another Zogenix-sponsored clinical trials with ZX008
* Subject's caregiver is willing and able to be compliant with study procedures, visit schedule and study drug accountability

Exclusion Criteria:

* Current cardiac valvulopathy or pulmonary hypertension that is clinically significant
* Moderate or severe hepatic impairment
* Receiving monoamine oxidase inhibitors, serotonin agonists, serotonin antagonists, and serotonin reuptake inhibitors within 14 days of receiving ZX008

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (71):
- United States (26):
  - Ep0215 107, Tucson, Arizona
  - Ep0215 144, Los Angeles, California
  - Ep0215 108, San Diego, California
  - Ep0215 101, San Francisco, California
  - Ep0215 103, Aurora, Colorado
  - Ep0215 115, Gulf Breeze, Florida
  - Ep0215 104, Miami, Florida
  - Ep0215 141, Orlando, Florida
  - Ep0215 121, Winter Park, Florida
  - Ep0215 117, Atlanta, Georgia
  - Ep0215 110, Chicago, Illinois
  - Ep0215 140, Bethesda, Maryland
  - Ep0215 112, Boston, Massachusetts
  - Ep0215 109, Rochester, Minnesota
  - Ep0215 132, Roseville, Minnesota
  - Ep0215 105, Hackensack, New Jersey
  - Ep0215 118, Livingston, New Jersey
  - Ep0215 150, Hawthorne, New York
  - Ep0215 142, New York, New York
  - Ep0215 131, Cleveland, Ohio
  - Ep0215 124, Memphis, Tennessee
  - Ep0215 146, Dallas, Texas
  - Ep0215 126, Fort Worth, Texas
  - Ep0215 106, Salt Lake City, Utah
  - Ep0215 119, Seattle, Washington
  - Ep0215 125, Tacoma, Washington
- Australia (3):
  - Ep0215 301, Heidelberg
  - Ep0215 302, South Brisbane
  - Ep0215 303, Westmead
- Belgium (3):
  - Ep0215 803, Brussels
  - Ep0215 801, Edegem
  - Ep0215 802, Jette
- Canada (3):
  - Ep0215 202, Montreal
  - Ep0215 204, Toronto
  - Ep0215 201, Vancouver
- Ep0215 701, Dianalund, Denmark
- France (6):
  - Ep0215 1004, Bordeaux
  - Ep0215 1005, Lille
  - Ep0215 1007, Marseille
  - Ep0215 1001, Paris
  - Ep0215 1002, Paris
  - Ep0215 1008, Salouël
- Germany (6):
  - Ep0215 902, Bielefeld
  - Ep0215 906, Freiburg im Breisgau
  - Ep0215 905, Jena
  - Ep0215 908, Kiel
  - Ep0215 903, Radeberg
  - Ep0215 901, Vogtareuth
- Italy (7):
  - Ep0215 1201, Florence
  - Ep0215 1204, Genova
  - Ep0215 1205, Mantova
  - Ep0215 1207, Milan
  - Ep0215 1206, Roma
  - Ep0215 1208, Roma
  - Ep0215 1202, Verona
- Ep0215 1604, Guadalajara, Mexico
- Netherlands (2):
  - Ep0215 1402, Heeze
  - Ep0215 1401, Zwolle
- Poland (2):
  - Ep0215 1702, Bydgoszcz
  - Ep0215 1701, Krakow
- Spain (5):
  - Ep0215 1105, Barcelona
  - Ep0215 1107, Barcelona
  - Ep0215 1103, Esplugues de Llobregat
  - Ep0215 1101, Madrid
  - Ep0215 1102, Pamplona
- Ep0215 502, Gothenburg, Sweden
- United Kingdom (5):
  - Ep0215 605, Birmingham
  - Ep0215 601, Glasgow
  - Ep0215 603, Liverpool
  - Ep0215 602, London
  - Ep0215 606, London

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://www.Vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in April 2019 and concluded in May 2025.
Pre-assignment Details: The Participant Flow refers to the Safety analysis set.
Groups:
- Any ZX008 Open Label Dose: Participants continued to receive ZX008 dose prescribed at last visit in ZX008-1503/EP0212 (NCT02823145), ZX008-1601/EP0214 Part 2 (NCT03355209), or ZX008-1602/EP0207 (NCT03467113) and had volume adjusted according to weight. In this Open Label Extension (OLE) study, participants who were not receiving concomitant Stiripentol (STP), dose could be titrated in increments of 0.2 mg/kg/day (milligram per kilogram per day) up to maximum of 0.8 mg/kg/day (not exceeding 30 mg/day). For participants receiving concomitant STP, dose could be adjusted to 0.4 mg/kg/day initially and increased to 0.5 mg/kg/day (not exceeding 20 mg/day). Participants continued ZX008 until one of following occurred: approval of ZX008 obtained from regulatory authorities for participants indication; managed access program established as per country-specific requirements, legal and regulatory guidelines in participants country of residence; or investigational product development for participants indication stopped by Sponsor.
Period: Overall Study
Arm/Group | Any ZX008 Open Label Dose
Started | 412
Completed | 360
Not Completed | 52
Not completed — Adverse Event | 3
Not completed — Death | 3
Not completed — Lack of Efficacy | 24
Not completed — Lost to Follow-up | 3
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 11
Not completed — Subjected Weaned of ZX008 | 1
Not completed — Missing | 6

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety analysis set which consisted of all participants who received at least one dose of ZX008 during the open label extension (OLE).
Arm/Group | Any ZX008 Open Label Dose
Number analyzed (Participants) | 412
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.1 (6.8)
Age, Customized [Count of Participants; unit: Participants]
  2 - <12 years | 168
  12 - <18 years | 117
  18 - <65 years | 127
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 191
  Male | 221
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 19
  Black or African American | 11
  Native Hawaiian or Other Pacific Islander | 1
  White | 327
  Other or Mixed | 4
  Not Reported | 35
  Unknown | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 60
  Not Hispanic or Latino | 303
  Not Reported | 42
  Unknown | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE can, therefore, be any unfavorable and unintended sign (including an abnormal, clinically significant laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product. TEAEs were defined as AE that began on or after the first day of treatment with ZX008 in Study EP0215 (ZX008-1900) (NCT03936777) or that occurred prior to first ZX008 treatment in Study EP0215 (ZX008-1900) but increased in severity after treatment in Study EP0215 (ZX008-1900) began. Events recorded at Follow-up/Cardiac Follow-up were considered treatment-emergent. The percentage of participants was rounded to one decimal place.
Time Frame: From First dose of ZX008 (in study EP0215 [ZX008-1900]) to Cardiac Follow-up after ZX008 treatment (Up to 6 Years, 17 Days)
Population: Safety analysis set consisted of participants who received at least one dose of ZX008 during the open label extension.
Measure: Number; unit: percentage of participants
Arm/Group | Any ZX008 Open Label Dose
Number analyzed (Participants) | 412
percentage of participants | 75.5

2. Secondary Outcome: Clinical Global Impression-Improvement in Participants, Subscale Global: Assessment by Parent/Caregiver
Description: The Clinical Global Impression-Improvement (CGI-I) scale is used to assess the severity of illness and global improvement in patients. Global function is one of the domains assessed by the CGI-I scale. The CGI-I is rated on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse) as follows: 1=Very much improved; 2=Much improved; 3=Minimally improved; 4=No change; 5=Minimally worse; 6=Much worse; 7=Very much worse, where higher score indicates worse outcome. The global CGI-I assessment was conducted by the Parent/Caregiver. The number of participants in each of the 7 categories of the CGI-I for each visit is reported.
Time Frame: Months 6, 12, 18, 24, 30, 36, Last On-Treatment Visit (Up to Month 49)
Population: The mITT analysis set consisted of all participants who received at least 1 dose of ZX008 and had at least one valid efficacy assessment during the OLE in the study EP0215 (ZX008-1900). Here, number of participants analyzed signifies participants who were evaluable for this outcome measure. Here, number analyzed signifies participants who were evaluable at specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Any ZX008 Open Label Dose
Number analyzed (Participants) | 401
Participants
  Month 6: Very much improved: number analyzed (Participants) | 371
  Month 6: Very much improved | 39
  Month 6: Much improved: number analyzed (Participants) | 371
  Month 6: Much improved | 88
  Month 6: Minimally improved: number analyzed (Participants) | 371
  Month 6: Minimally improved | 87
  Month 6: No change: number analyzed (Participants) | 371
  Month 6: No change | 124
  Month 6: Minimally worse: number analyzed (Participants) | 371
  Month 6: Minimally worse | 23
  Month 6: Much worse: number analyzed (Participants) | 371
  Month 6: Much worse | 7
  Month 6: Very much worse: number analyzed (Participants) | 371
  Month 6: Very much worse | 3
  Month 12: Very much improved: number analyzed (Participants) | 266
  Month 12: Very much improved | 42
  Month 12: Much improved: number analyzed (Participants) | 266
  Month 12: Much improved | 65
  Month 12: Minimally improved: number analyzed (Participants) | 266
  Month 12: Minimally improved | 56
  Month 12: No change: number analyzed (Participants) | 266
  Month 12: No change | 77
  Month 12: Minimally worse: number analyzed (Participants) | 266
  Month 12: Minimally worse | 17
  Month 12: Much worse: number analyzed (Participants) | 266
  Month 12: Much worse | 9
  Month 12: Very much worse: number analyzed (Participants) | 266
  Month 12: Very much worse | 0
  Month 18: Very much improved: number analyzed (Participants) | 223
  Month 18: Very much improved | 34
  Month 18: Much improved: number analyzed (Participants) | 223
  Month 18: Much improved | 43
  Month 18: Minimally improved: number analyzed (Participants) | 223
  Month 18: Minimally improved | 60
  Month 18: No change: number analyzed (Participants) | 223
  Month 18: No change | 67
  Month 18: Minimally worse: number analyzed (Participants) | 223
  Month 18: Minimally worse | 16
  Month 18: Much worse: number analyzed (Participants) | 223
  Month 18: Much worse | 2
  Month 18: Very much worse: number analyzed (Participants) | 223
  Month 18: Very much worse | 1
  Month 24: Very much improved: number analyzed (Participants) | 188
  Month 24: Very much improved | 33
  Month 24: Much improved: number analyzed (Participants) | 188
  Month 24: Much improved | 46
  Month 24: Minimally improved: number analyzed (Participants) | 188
  Month 24: Minimally improved | 41
  Month 24: No change: number analyzed (Participants) | 188
  Month 24: No change | 59
  Month 24: Minimally worse: number analyzed (Participants) | 188
  Month 24: Minimally worse | 8
  Month 24: Much worse: number analyzed (Participants) | 188
  Month 24: Much worse | 1
  Month 24: Very much worse: number analyzed (Participants) | 188
  Month 24: Very much worse | 0
  Month 30: Very much improved: number analyzed (Participants) | 149
  Month 30: Very much improved | 16
  Month 30: Much improved: number analyzed (Participants) | 149
  Month 30: Much improved | 41
  Month 30: Minimally improved: number analyzed (Participants) | 149
  Month 30: Minimally improved | 34
  Month 30: No change: number analyzed (Participants) | 149
  Month 30: No change | 47
  Month 30: Minimally worse: number analyzed (Participants) | 149
  Month 30: Minimally worse | 9
  Month 30: Much worse: number analyzed (Participants) | 149
  Month 30: Much worse | 1
  Month 30: Very much worse: number analyzed (Participants) | 149
  Month 30: Very much worse | 1
  Month 36: Very much improved: number analyzed (Participants) | 128
  Month 36: Very much improved | 16
  Month 36: Much improved: number analyzed (Participants) | 128
  Month 36: Much improved | 31
  Month 36: Minimally improved: number analyzed (Participants) | 128
  Month 36: Minimally improved | 29
  Month 36: No change: number analyzed (Participants) | 128
  Month 36: No change | 39
  Month 36: Minimally worse: number analyzed (Participants) | 128
  Month 36: Minimally worse | 10
  Month 36: Much worse: number analyzed (Participants) | 128
  Month 36: Much worse | 3
  Month 36: Very much worse: number analyzed (Participants) | 128
  Month 36: Very much worse | 0
  Last On-Treatment Visit: Very much improved | 71
  Last On-Treatment Visit: Much improved | 109
  Last On-Treatment Visit: Minimally improved | 85
  Last On-Treatment Visit: No change | 108
  Last On-Treatment Visit: Minimally worse | 21
  Last On-Treatment Visit: Much worse | 7
  Last On-Treatment Visit: Very much worse | 0

3. Secondary Outcome: Clinical Global Impression-Improvement in Participants, Subscale Global: Assessment by Investigator
Description: The CGI-I scale is used to assess the severity of illness and global improvement in patients. Global function is one of the domains assessed by the CGI-I scale. The CGI-I is rated on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse) as follows: 1=Very much improved; 2=Much improved; 3=Minimally improved; 4=No change; 5=Minimally worse; 6=Much worse; 7=Very much worse, where higher score indicates worse outcome. The global CGI-I assessment was conducted by the Investigator. The number of participants in each of the 7 categories of the CGI-I for each visit is reported.
Time Frame: Months 6, 12, 18, 24, 30, 36, Last On-Treatment Visit (Up to Month 49)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Any ZX008 Open Label Dose
Number analyzed (Participants) | 401
Participants
  Month 6: Very much improved: number analyzed (Participants) | 367
  Month 6: Very much improved | 23
  Month 6: Much improved: number analyzed (Participants) | 367
  Month 6: Much improved | 86
  Month 6: Minimally improved: number analyzed (Participants) | 367
  Month 6: Minimally improved | 85
  Month 6: No change: number analyzed (Participants) | 367
  Month 6: No change | 141
  Month 6: Minimally worse: number analyzed (Participants) | 367
  Month 6: Minimally worse | 26
  Month 6: Much worse: number analyzed (Participants) | 367
  Month 6: Much worse | 4
  Month 6: Very much worse: number analyzed (Participants) | 367
  Month 6: Very much worse | 2
  Month 12: Very much improved: number analyzed (Participants) | 265
  Month 12: Very much improved | 28
  Month 12: Much improved: number analyzed (Participants) | 265
  Month 12: Much improved | 63
  Month 12: Minimally improved: number analyzed (Participants) | 265
  Month 12: Minimally improved | 66
  Month 12: No change: number analyzed (Participants) | 265
  Month 12: No change | 87
  Month 12: Minimally worse: number analyzed (Participants) | 265
  Month 12: Minimally worse | 17
  Month 12: Much worse: number analyzed (Participants) | 265
  Month 12: Much worse | 3
  Month 12: Very much worse: number analyzed (Participants) | 265
  Month 12: Very much worse | 1
  Month 18: Very much improved: number analyzed (Participants) | 225
  Month 18: Very much improved | 23
  Month 18: Much improved: number analyzed (Participants) | 225
  Month 18: Much improved | 45
  Month 18: Minimally improved: number analyzed (Participants) | 225
  Month 18: Minimally improved | 58
  Month 18: No change: number analyzed (Participants) | 225
  Month 18: No change | 86
  Month 18: Minimally worse: number analyzed (Participants) | 225
  Month 18: Minimally worse | 12
  Month 18: Much worse: number analyzed (Participants) | 225
  Month 18: Much worse | 1
  Month 18: Very much worse: number analyzed (Participants) | 225
  Month 18: Very much worse | 0
  Month 24: Very much improved: number analyzed (Participants) | 189
  Month 24: Very much improved | 20
  Month 24: Much improved: number analyzed (Participants) | 189
  Month 24: Much improved | 54
  Month 24: Minimally improved: number analyzed (Participants) | 189
  Month 24: Minimally improved | 37
  Month 24: No change: number analyzed (Participants) | 189
  Month 24: No change | 72
  Month 24: Minimally worse: number analyzed (Participants) | 189
  Month 24: Minimally worse | 5
  Month 24: Much worse: number analyzed (Participants) | 189
  Month 24: Much worse | 1
  Month 24: Very much worse: number analyzed (Participants) | 189
  Month 24: Very much worse | 0
  Month 30: Very much improved: number analyzed (Participants) | 149
  Month 30: Very much improved | 11
  Month 30: Much improved: number analyzed (Participants) | 149
  Month 30: Much improved | 44
  Month 30: Minimally improved: number analyzed (Participants) | 149
  Month 30: Minimally improved | 34
  Month 30: No change: number analyzed (Participants) | 149
  Month 30: No change | 56
  Month 30: Minimally worse: number analyzed (Participants) | 149
  Month 30: Minimally worse | 3
  Month 30: Much worse: number analyzed (Participants) | 149
  Month 30: Much worse | 1
  Month 30: Very much worse: number analyzed (Participants) | 149
  Month 30: Very much worse | 0
  Month 36: Very much improved: number analyzed (Participants) | 124
  Month 36: Very much improved | 7
  Month 36: Much improved: number analyzed (Participants) | 124
  Month 36: Much improved | 33
  Month 36: Minimally improved: number analyzed (Participants) | 124
  Month 36: Minimally improved | 25
  Month 36: No change: number analyzed (Participants) | 124
  Month 36: No change | 52
  Month 36: Minimally worse: number analyzed (Participants) | 124
  Month 36: Minimally worse | 5
  Month 36: Much worse: number analyzed (Participants) | 124
  Month 36: Much worse | 2
  Month 36: Very much worse: number analyzed (Participants) | 124
  Month 36: Very much worse | 0
  Last On-Treatment Visit: Very much improved | 33
  Last On-Treatment Visit: Much improved | 108
  Last On-Treatment Visit: Minimally improved | 101
  Last On-Treatment Visit: No change | 134
  Last On-Treatment Visit: Minimally worse | 19
  Last On-Treatment Visit: Much worse | 5
  Last On-Treatment Visit: Very much worse | 1

4. Secondary Outcome: Clinical Global Impression-Improvement in Participants, Subscale Cognition: Assessment by Parent/Caregiver
Description: The CGI-I scale is used to assess the severity of illness and global improvement in patients. Cognitive function is one of the domains assessed by the CGI-I scale. The CGI-I is rated on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse) as follows: 1=Very much improved; 2=Much improved; 3=Minimally improved; 4=No change; 5=Minimally worse; 6=Much worse; 7=Very much worse, where higher score indicates worse outcome. The CGI-I assessment of cognition was conducted by the Parent/Caregiver. The number of participants in each of the 7 categories of the CGI-I for each visit is reported.
Time Frame: Months 6, 12, 18, 24, 30, 36, Last On-Treatment Visit (Up to Month 49)
Population: The modified Intent-to-Treat (mITT) analysis set consisted of all participants who received at least 1 dose of ZX008 and had at least one valid efficacy assessment during the open-label extension (OLE) in the study EP0215 (ZX008-1900). Here, number of participants analyzed signifies participants who were evaluable for this outcome measure. Here, number analyzed signifies participants who were evaluable at specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Any ZX008 Open Label Dose
Number analyzed (Participants) | 401
Participants
  Month 6: Very much improved: number analyzed (Participants) | 370
  Month 6: Very much improved | 26 [4.6 to 10.1]
  Month 6: Much improved: number analyzed (Participants) | 370
  Month 6: Much improved | 75 [16.3 to 24.7]
  Month 6: Minimally improved: number analyzed (Participants) | 370
  Month 6: Minimally improved | 87 [19.3 to 28.2]
  Month 6: No change: number analyzed (Participants) | 370
  Month 6: No change | 161 [38.4 to 48.7]
  Month 6: Minimally worse: number analyzed (Participants) | 370
  Month 6: Minimally worse | 15 [2.3 to 6.6]
  Month 6: Much worse: number analyzed (Participants) | 370
  Month 6: Much worse | 4 [0.3 to 2.7]
  Month 6: Very much worse: number analyzed (Participants) | 370
  Month 6: Very much worse | 2 [0.1 to 1.9]
  Month 12: Very much improved: number analyzed (Participants) | 265
  Month 12: Very much improved | 17 [3.8 to 10.1]
  Month 12: Much improved: number analyzed (Participants) | 265
  Month 12: Much improved | 54 [15.7 to 25.7]
  Month 12: Minimally improved: number analyzed (Participants) | 265
  Month 12: Minimally improved | 78 [24.0 to 35.3]
  Month 12: No change: number analyzed (Participants) | 265
  Month 12: No change | 108 [34.8 to 46.9]
  Month 12: Minimally worse: number analyzed (Participants) | 265
  Month 12: Minimally worse | 5 [0.6 to 4.3]
  Month 12: Much worse: number analyzed (Participants) | 265
  Month 12: Much worse | 3 [0.2 to 3.3]
  Month 12: Very much worse: number analyzed (Participants) | 265
  Month 12: Very much worse | 0 [0 to 1.4]
  Month 18: Very much improved: number analyzed (Participants) | 224
  Month 18: Very much improved | 18 [4.8 to 12.4]
  Month 18: Much improved: number analyzed (Participants) | 224
  Month 18: Much improved | 43 [14.3 to 25.0]
  Month 18: Minimally improved: number analyzed (Participants) | 224
  Month 18: Minimally improved | 69 [24.8 to 37.3]
  Month 18: No change: number analyzed (Participants) | 224
  Month 18: No change | 86 [32.0 to 45.1]
  Month 18: Minimally worse: number analyzed (Participants) | 224
  Month 18: Minimally worse | 6 [1.0 to 5.7]
  Month 18: Much worse: number analyzed (Participants) | 224
  Month 18: Much worse | 2 [0.1 to 3.2]
  Month 18: Very much worse: number analyzed (Participants) | 224
  Month 18: Very much worse | 0 [0 to 1.6]
  Month 24: Very much improved: number analyzed (Participants) | 188
  Month 24: Very much improved | 14 [4.1 to 12.2]
  Month 24: Much improved: number analyzed (Participants) | 188
  Month 24: Much improved | 35 [13.3 to 24.9]
  Month 24: Minimally improved: number analyzed (Participants) | 188
  Month 24: Minimally improved | 59 [24.8 to 38.5]
  Month 24: No change: number analyzed (Participants) | 188
  Month 24: No change | 73 [31.8 to 46.2]
  Month 24: Minimally worse: number analyzed (Participants) | 188
  Month 24: Minimally worse | 6 [1.2 to 6.8]
  Month 24: Much worse: number analyzed (Participants) | 188
  Month 24: Much worse | 1 [0.0 to 2.9]
  Month 24: Very much worse: number analyzed (Participants) | 188
  Month 24: Very much worse | 0 [0 to 1.9]
  Month 30: Very much improved: number analyzed (Participants) | 149
  Month 30: Very much improved | 7 [1.9 to 9.4]
  Month 30: Much improved: number analyzed (Participants) | 149
  Month 30: Much improved | 31 [14.6 to 28.2]
  Month 30: Minimally improved: number analyzed (Participants) | 149
  Month 30: Minimally improved | 41 [20.5 to 35.4]
  Month 30: No change: number analyzed (Participants) | 149
  Month 30: No change | 62 [33.6 to 50.0]
  Month 30: Minimally worse: number analyzed (Participants) | 149
  Month 30: Minimally worse | 6 [1.5 to 8.6]
  Month 30: Much worse: number analyzed (Participants) | 149
  Month 30: Much worse | 1 [0.0 to 3.7]
  Month 30: Very much worse: number analyzed (Participants) | 149
  Month 30: Very much worse | 1 [0.0 to 3.7]
  Month 36: Very much improved: number analyzed (Participants) | 128
  Month 36: Very much improved | 6 [1.7 to 9.9]
  Month 36: Much improved: number analyzed (Participants) | 128
  Month 36: Much improved | 32 [17.8 to 33.4]
  Month 36: Minimally improved: number analyzed (Participants) | 128
  Month 36: Minimally improved | 29 [15.7 to 30.9]
  Month 36: No change: number analyzed (Participants) | 128
  Month 36: No change | 49 [29.8 to 47.3]
  Month 36: Minimally worse: number analyzed (Participants) | 128
  Month 36: Minimally worse | 11 [4.4 to 14.9]
  Month 36: Much worse: number analyzed (Participants) | 128
  Month 36: Much worse | 1 [0.0 to 4.3]
  Month 36: Very much worse: number analyzed (Participants) | 128
  Month 36: Very much worse | 0 [0 to 2.8]
  Last On-Treatment Visit: Very much improved | 33 [5.7 to 11.4]
  Last On-Treatment Visit: Much improved | 98 [20.3 to 28.9]
  Last On-Treatment Visit: Minimally improved | 101 [21.0 to 29.7]
  Last On-Treatment Visit: No change | 148 [32.2 to 41.8]
  Last On-Treatment Visit: Minimally worse | 16 [2.3 to 6.4]
  Last On-Treatment Visit: Much worse | 5 [0.4 to 2.9]
  Last On-Treatment Visit: Very much worse | 0 [0 to 0.9]

5. Secondary Outcome: Clinical Global Impression-Improvement in Participants, Subscale Behavior: Assessment by Parent/Caregiver
Description: The CGI-I scale is used to assess the severity of illness and global improvement in patients. Behavior is one of the domains assessed by the CGI-I scale. The CGI-I is rated on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse) as follows: 1=Very much improved; 2=Much improved; 3=Minimally improved; 4=No change; 5=Minimally worse; 6=Much worse; 7=Very much worse, where higher score indicates worse outcome. The CGI-I assessment of behavior was conducted by the Parent/Caregiver. The number of participants in each of the 7 categories of the CGI-I for each visit is reported.
Time Frame: Months 6, 12, 18, 24, 30, 36, Last On-Treatment Visit (Up to Month 49)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Any ZX008 Open Label Dose
Number analyzed (Participants) | 401
Participants
  Month 6: Very much improved: number analyzed (Participants) | 370
  Month 6: Very much improved | 20
  Month 6: Much improved: number analyzed (Participants) | 370
  Month 6: Much improved | 51
  Month 6: Minimally improved: number analyzed (Participants) | 370
  Month 6: Minimally improved | 75
  Month 6: No change: number analyzed (Participants) | 370
  Month 6: No change | 174
  Month 6: Minimally worse: number analyzed (Participants) | 370
  Month 6: Minimally worse | 35
  Month 6: Much worse: number analyzed (Participants) | 370
  Month 6: Much worse | 12
  Month 6: Very much worse: number analyzed (Participants) | 370
  Month 6: Very much worse | 3
  Month 12: Very much improved: number analyzed (Participants) | 265
  Month 12: Very much improved | 9
  Month 12: Much improved: number analyzed (Participants) | 265
  Month 12: Much improved | 46
  Month 12: Minimally improved: number analyzed (Participants) | 265
  Month 12: Minimally improved | 51
  Month 12: No change: number analyzed (Participants) | 265
  Month 12: No change | 120
  Month 12: Minimally worse: number analyzed (Participants) | 265
  Month 12: Minimally worse | 28
  Month 12: Much worse: number analyzed (Participants) | 265
  Month 12: Much worse | 11
  Month 12: Very much worse: number analyzed (Participants) | 265
  Month 12: Very much worse | 0
  Month 18: Very much improved: number analyzed (Participants) | 224
  Month 18: Very much improved | 13
  Month 18: Much improved: number analyzed (Participants) | 224
  Month 18: Much improved | 37
  Month 18: Minimally improved: number analyzed (Participants) | 224
  Month 18: Minimally improved | 42
  Month 18: No change: number analyzed (Participants) | 224
  Month 18: No change | 100
  Month 18: Minimally worse: number analyzed (Participants) | 224
  Month 18: Minimally worse | 27
  Month 18: Much worse: number analyzed (Participants) | 224
  Month 18: Much worse | 4
  Month 18: Very much worse: number analyzed (Participants) | 224
  Month 18: Very much worse | 1
  Month 24: Very much improved: number analyzed (Participants) | 188
  Month 24: Very much improved | 13
  Month 24: Much improved: number analyzed (Participants) | 188
  Month 24: Much improved | 31
  Month 24: Minimally improved: number analyzed (Participants) | 188
  Month 24: Minimally improved | 36
  Month 24: No change: number analyzed (Participants) | 188
  Month 24: No change | 83
  Month 24: Minimally worse: number analyzed (Participants) | 188
  Month 24: Minimally worse | 16
  Month 24: Much worse: number analyzed (Participants) | 188
  Month 24: Much worse | 9
  Month 24: Very much worse: number analyzed (Participants) | 188
  Month 24: Very much worse | 0
  Month 30: Very much improved: number analyzed (Participants) | 149
  Month 30: Very much improved | 8
  Month 30: Much improved: number analyzed (Participants) | 149
  Month 30: Much improved | 26
  Month 30: Minimally improved: number analyzed (Participants) | 149
  Month 30: Minimally improved | 27
  Month 30: No change: number analyzed (Participants) | 149
  Month 30: No change | 69
  Month 30: Minimally worse: number analyzed (Participants) | 149
  Month 30: Minimally worse | 15
  Month 30: Much worse: number analyzed (Participants) | 149
  Month 30: Much worse | 4
  Month 30: Very much worse: number analyzed (Participants) | 149
  Month 30: Very much worse | 0
  Month 36: Very much improved: number analyzed (Participants) | 128
  Month 36: Very much improved | 7
  Month 36: Much improved: number analyzed (Participants) | 128
  Month 36: Much improved | 18
  Month 36: Minimally improved: number analyzed (Participants) | 128
  Month 36: Minimally improved | 28
  Month 36: No change: number analyzed (Participants) | 128
  Month 36: No change | 58
  Month 36: Minimally worse: number analyzed (Participants) | 128
  Month 36: Minimally worse | 10
  Month 36: Much worse: number analyzed (Participants) | 128
  Month 36: Much worse | 6
  Month 36: Very much worse: number analyzed (Participants) | 128
  Month 36: Very much worse | 1
  Last On-Treatment Visit: Very much improved | 24
  Last On-Treatment Visit: Much improved | 73
  Last On-Treatment Visit: Minimally improved | 83
  Last On-Treatment Visit: No change | 169
  Last On-Treatment Visit: Minimally worse | 36
  Last On-Treatment Visit: Much worse | 15
  Last On-Treatment Visit: Very much worse | 1

6. Secondary Outcome: Clinical Global Impression-Improvement in Participants, Subscale Motor Abilities: Assessment by Parent/Caregiver
Description: The CGI-I scale is used to assess the severity of illness and global improvement in patients. Motor abilities function is one of the domains assessed by the CGI-I scale. The CGI-I is rated on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse) as follows: 1=Very much improved; 2=Much improved; 3=Minimally improved; 4=No change; 5=Minimally worse; 6=Much worse; 7=Very much worse, where higher score indicates worse outcome. The CGI-I assessment of motor abilities was conducted by the Parent/Caregiver. The number of participants in each of the 7 categories of the CGI-I for each visit is reported.
Time Frame: Months 6, 12, 18, 24, 30, 36, Last On-Treatment Visit (Up to Month 49)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Any ZX008 Open Label Dose
Number analyzed (Participants) | 401
Participants
  Month 6: Very much improved: number analyzed (Participants) | 370
  Month 6: Very much improved | 17
  Month 6: Much improved: number analyzed (Participants) | 370
  Month 6: Much improved | 45
  Month 6: Minimally improved: number analyzed (Participants) | 370
  Month 6: Minimally improved | 86
  Month 6: No change: number analyzed (Participants) | 370
  Month 6: No change | 190
  Month 6: Minimally worse: number analyzed (Participants) | 370
  Month 6: Minimally worse | 26
  Month 6: Much worse: number analyzed (Participants) | 370
  Month 6: Much worse | 4
  Month 6: Very much worse: number analyzed (Participants) | 370
  Month 6: Very much worse | 2
  Month 12: Very much improved: number analyzed (Participants) | 265
  Month 12: Very much improved | 14
  Month 12: Much improved: number analyzed (Participants) | 265
  Month 12: Much improved | 31
  Month 12: Minimally improved: number analyzed (Participants) | 265
  Month 12: Minimally improved | 65
  Month 12: No change: number analyzed (Participants) | 265
  Month 12: No change | 134
  Month 12: Minimally worse: number analyzed (Participants) | 265
  Month 12: Minimally worse | 14
  Month 12: Much worse: number analyzed (Participants) | 265
  Month 12: Much worse | 6
  Month 12: Very much worse: number analyzed (Participants) | 265
  Month 12: Very much worse | 1
  Month 18: Very much improved: number analyzed (Participants) | 224
  Month 18: Very much improved | 10
  Month 18: Much improved: number analyzed (Participants) | 224
  Month 18: Much improved | 31
  Month 18: Minimally improved: number analyzed (Participants) | 224
  Month 18: Minimally improved | 48
  Month 18: No change: number analyzed (Participants) | 224
  Month 18: No change | 114
  Month 18: Minimally worse: number analyzed (Participants) | 224
  Month 18: Minimally worse | 16
  Month 18: Much worse: number analyzed (Participants) | 224
  Month 18: Much worse | 4
  Month 18: Very much worse: number analyzed (Participants) | 224
  Month 18: Very much worse | 1
  Month 24: Very much improved: number analyzed (Participants) | 188
  Month 24: Very much improved | 16
  Month 24: Much improved: number analyzed (Participants) | 188
  Month 24: Much improved | 19
  Month 24: Minimally improved: number analyzed (Participants) | 188
  Month 24: Minimally improved | 42
  Month 24: No change: number analyzed (Participants) | 188
  Month 24: No change | 97
  Month 24: Minimally worse: number analyzed (Participants) | 188
  Month 24: Minimally worse | 13
  Month 24: Much worse: number analyzed (Participants) | 188
  Month 24: Much worse | 1
  Month 24: Very much worse: number analyzed (Participants) | 188
  Month 24: Very much worse | 0
  Month 30: Very much improved: number analyzed (Participants) | 149
  Month 30: Very much improved | 7
  Month 30: Much improved: number analyzed (Participants) | 149
  Month 30: Much improved | 22
  Month 30: Minimally improved: number analyzed (Participants) | 149
  Month 30: Minimally improved | 27
  Month 30: No change: number analyzed (Participants) | 149
  Month 30: No change | 77
  Month 30: Minimally worse: number analyzed (Participants) | 149
  Month 30: Minimally worse | 13
  Month 30: Much worse: number analyzed (Participants) | 149
  Month 30: Much worse | 2
  Month 30: Very much worse: number analyzed (Participants) | 149
  Month 30: Very much worse | 1
  Month 36: Very much improved: number analyzed (Participants) | 128
  Month 36: Very much improved | 6
  Month 36: Much improved: number analyzed (Participants) | 128
  Month 36: Much improved | 16
  Month 36: Minimally improved: number analyzed (Participants) | 128
  Month 36: Minimally improved | 22
  Month 36: No change: number analyzed (Participants) | 128
  Month 36: No change | 67
  Month 36: Minimally worse: number analyzed (Participants) | 128
  Month 36: Minimally worse | 9
  Month 36: Much worse: number analyzed (Participants) | 128
  Month 36: Much worse | 7
  Month 36: Very much worse: number analyzed (Participants) | 128
  Month 36: Very much worse | 1
  Last On-Treatment Visit: Very much improved | 24
  Last On-Treatment Visit: Much improved | 55
  Last On-Treatment Visit: Minimally improved | 94
  Last On-Treatment Visit: No change | 191
  Last On-Treatment Visit: Minimally worse | 25
  Last On-Treatment Visit: Much worse | 12
  Last On-Treatment Visit: Very much worse | 0

7. Secondary Outcome: Clinical Global Impression-Improvement in Participants, Subscale Cognition: Assessment by Investigator
Description: The CGI-I scale is used to assess the severity of illness and global improvement in patients. Cognitive function is one of the domains assessed by the CGI-I scale. The CGI-I is rated on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse) as follows: 1=Very much improved; 2=Much improved; 3=Minimally improved; 4=No change; 5=Minimally worse; 6=Much worse; 7=Very much worse, where higher score indicates worse outcome. The CGI-I assessment of cognition was conducted by the Investigator. The number of participants in each of the 7 categories of the CGI-I for each visit is reported.
Time Frame: Months 6, 12, 18, 24, 30, 36, Last On-Treatment Visit (Up to Month 49)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Any ZX008 Open Label Dose
Number analyzed (Participants) | 399
Participants
  Month 6: Very much improved: number analyzed (Participants) | 365
  Month 6: Very much improved | 13
  Month 6: Much improved: number analyzed (Participants) | 365
  Month 6: Much improved | 54
  Month 6: Minimally improved: number analyzed (Participants) | 365
  Month 6: Minimally improved | 101
  Month 6: No change: number analyzed (Participants) | 365
  Month 6: No change | 184
  Month 6: Minimally worse: number analyzed (Participants) | 365
  Month 6: Minimally worse | 9
  Month 6: Much worse: number analyzed (Participants) | 365
  Month 6: Much worse | 2
  Month 6: Very much worse: number analyzed (Participants) | 365
  Month 6: Very much worse | 2
  Month 12: Very much improved: number analyzed (Participants) | 265
  Month 12: Very much improved | 13
  Month 12: Much improved: number analyzed (Participants) | 265
  Month 12: Much improved | 39
  Month 12: Minimally improved: number analyzed (Participants) | 265
  Month 12: Minimally improved | 79
  Month 12: No change: number analyzed (Participants) | 265
  Month 12: No change | 128
  Month 12: Minimally worse: number analyzed (Participants) | 265
  Month 12: Minimally worse | 4
  Month 12: Much worse: number analyzed (Participants) | 265
  Month 12: Much worse | 1
  Month 12: Very much worse: number analyzed (Participants) | 265
  Month 12: Very much worse | 1
  Month 18: Very much improved: number analyzed (Participants) | 226
  Month 18: Very much improved | 13
  Month 18: Much improved: number analyzed (Participants) | 226
  Month 18: Much improved | 32
  Month 18: Minimally improved: number analyzed (Participants) | 226
  Month 18: Minimally improved | 53
  Month 18: No change: number analyzed (Participants) | 226
  Month 18: No change | 118
  Month 18: Minimally worse: number analyzed (Participants) | 226
  Month 18: Minimally worse | 10
  Month 18: Much worse: number analyzed (Participants) | 226
  Month 18: Much worse | 0
  Month 18: Very much worse: number analyzed (Participants) | 226
  Month 18: Very much worse | 0
  Month 24: Very much improved: number analyzed (Participants) | 189
  Month 24: Very much improved | 9
  Month 24: Much improved: number analyzed (Participants) | 189
  Month 24: Much improved | 33
  Month 24: Minimally improved: number analyzed (Participants) | 189
  Month 24: Minimally improved | 55
  Month 24: No change: number analyzed (Participants) | 189
  Month 24: No change | 88
  Month 24: Minimally worse: number analyzed (Participants) | 189
  Month 24: Minimally worse | 3
  Month 24: Much worse: number analyzed (Participants) | 189
  Month 24: Much worse | 1
  Month 24: Very much worse: number analyzed (Participants) | 189
  Month 24: Very much worse | 0
  Month 30: Very much improved: number analyzed (Participants) | 149
  Month 30: Very much improved | 4
  Month 30: Much improved: number analyzed (Participants) | 149
  Month 30: Much improved | 25
  Month 30: Minimally improved: number analyzed (Participants) | 149
  Month 30: Minimally improved | 36
  Month 30: No change: number analyzed (Participants) | 149
  Month 30: No change | 81
  Month 30: Minimally worse: number analyzed (Participants) | 149
  Month 30: Minimally worse | 3
  Month 30: Much worse: number analyzed (Participants) | 149
  Month 30: Much worse | 0
  Month 30: Very much worse: number analyzed (Participants) | 149
  Month 30: Very much worse | 0
  Month 36: Very much improved: number analyzed (Participants) | 124
  Month 36: Very much improved | 4
  Month 36: Much improved: number analyzed (Participants) | 124
  Month 36: Much improved | 14
  Month 36: Minimally improved: number analyzed (Participants) | 124
  Month 36: Minimally improved | 34
  Month 36: No change: number analyzed (Participants) | 124
  Month 36: No change | 65
  Month 36: Minimally worse: number analyzed (Participants) | 124
  Month 36: Minimally worse | 7
  Month 36: Much worse: number analyzed (Participants) | 124
  Month 36: Much worse | 0
  Month 36: Very much worse: number analyzed (Participants) | 124
  Month 36: Very much worse | 0
  Last On-Treatment Visit: Very much improved | 16
  Last On-Treatment Visit: Much improved | 64
  Last On-Treatment Visit: Minimally improved | 103
  Last On-Treatment Visit: No change | 201
  Last On-Treatment Visit: Minimally worse | 12
  Last On-Treatment Visit: Much worse | 1
  Last On-Treatment Visit: Very much worse | 2

8. Secondary Outcome: Clinical Global Impression-Improvement in Participants, Subscale Behavior: Assessment by Investigator
Description: The CGI-I scale is used to assess the severity of illness and global improvement in patients. Behavior is one of the domains assessed by the CGI-I scale. The CGI-I is rated on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse) as follows: 1=Very much improved; 2=Much improved; 3=Minimally improved; 4=No change; 5=Minimally worse; 6=Much worse; 7=Very much worse, where higher score indicates worse outcome. The CGI-I assessment of behavior was conducted by the Investigator. The number of participants in each of the 7 categories of the CGI-I for each visit is reported.
Time Frame: Months 6, 12, 18, 24, 30, 36, Last On-Treatment Visit (Up to Month 49)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Any ZX008 Open Label Dose
Number analyzed (Participants) | 399
Participants
  Month 6: Very much improved: number analyzed (Participants) | 365
  Month 6: Very much improved | 10
  Month 6: Much improved: number analyzed (Participants) | 365
  Month 6: Much improved | 42
  Month 6: Minimally improved: number analyzed (Participants) | 365
  Month 6: Minimally improved | 80
  Month 6: No change: number analyzed (Participants) | 365
  Month 6: No change | 200
  Month 6: Minimally worse: number analyzed (Participants) | 365
  Month 6: Minimally worse | 27
  Month 6: Much worse: number analyzed (Participants) | 365
  Month 6: Much worse | 5
  Month 6: Very much worse: number analyzed (Participants) | 365
  Month 6: Very much worse | 1
  Month 12: Very much improved: number analyzed (Participants) | 265
  Month 12: Very much improved | 11
  Month 12: Much improved: number analyzed (Participants) | 265
  Month 12: Much improved | 35
  Month 12: Minimally improved: number analyzed (Participants) | 265
  Month 12: Minimally improved | 54
  Month 12: No change: number analyzed (Participants) | 265
  Month 12: No change | 144
  Month 12: Minimally worse: number analyzed (Participants) | 265
  Month 12: Minimally worse | 17
  Month 12: Much worse: number analyzed (Participants) | 265
  Month 12: Much worse | 3
  Month 12: Very much worse: number analyzed (Participants) | 265
  Month 12: Very much worse | 1
  Month 18: Very much improved: number analyzed (Participants) | 226
  Month 18: Very much improved | 7
  Month 18: Much improved: number analyzed (Participants) | 226
  Month 18: Much improved | 32
  Month 18: Minimally improved: number analyzed (Participants) | 226
  Month 18: Minimally improved | 41
  Month 18: No change: number analyzed (Participants) | 226
  Month 18: No change | 122
  Month 18: Minimally worse: number analyzed (Participants) | 226
  Month 18: Minimally worse | 20
  Month 18: Much worse: number analyzed (Participants) | 226
  Month 18: Much worse | 3
  Month 18: Very much worse: number analyzed (Participants) | 226
  Month 18: Very much worse | 1
  Month 24: Very much improved: number analyzed (Participants) | 189
  Month 24: Very much improved | 11
  Month 24: Much improved: number analyzed (Participants) | 189
  Month 24: Much improved | 28
  Month 24: Minimally improved: number analyzed (Participants) | 189
  Month 24: Minimally improved | 36
  Month 24: No change: number analyzed (Participants) | 189
  Month 24: No change | 95
  Month 24: Minimally worse: number analyzed (Participants) | 189
  Month 24: Minimally worse | 17
  Month 24: Much worse: number analyzed (Participants) | 189
  Month 24: Much worse | 2
  Month 24: Very much worse: number analyzed (Participants) | 189
  Month 24: Very much worse | 0
  Month 30: Very much improved: number analyzed (Participants) | 149
  Month 30: Very much improved | 2
  Month 30: Much improved: number analyzed (Participants) | 149
  Month 30: Much improved | 28
  Month 30: Minimally improved: number analyzed (Participants) | 149
  Month 30: Minimally improved | 25
  Month 30: No change: number analyzed (Participants) | 149
  Month 30: No change | 77
  Month 30: Minimally worse: number analyzed (Participants) | 149
  Month 30: Minimally worse | 15
  Month 30: Much worse: number analyzed (Participants) | 149
  Month 30: Much worse | 2
  Month 30: Very much worse: number analyzed (Participants) | 149
  Month 30: Very much worse | 0
  Month 36: Very much improved: number analyzed (Participants) | 124
  Month 36: Very much improved | 1
  Month 36: Much improved: number analyzed (Participants) | 124
  Month 36: Much improved | 19
  Month 36: Minimally improved: number analyzed (Participants) | 124
  Month 36: Minimally improved | 28
  Month 36: No change: number analyzed (Participants) | 124
  Month 36: No change | 63
  Month 36: Minimally worse: number analyzed (Participants) | 124
  Month 36: Minimally worse | 11
  Month 36: Much worse: number analyzed (Participants) | 124
  Month 36: Much worse | 2
  Month 36: Very much worse: number analyzed (Participants) | 124
  Month 36: Very much worse | 0
  Last On-Treatment Visit: Very much improved | 14
  Last On-Treatment Visit: Much improved | 57
  Last On-Treatment Visit: Minimally improved | 74
  Last On-Treatment Visit: No change | 229
  Last On-Treatment Visit: Minimally worse | 20
  Last On-Treatment Visit: Much worse | 3
  Last On-Treatment Visit: Very much worse | 2

9. Secondary Outcome: Clinical Global Impression Improvement in Participants, Subscale Motor Abilities: Assessment by Investigator
Description: The CGI-I scale is used to assess the severity of illness and global improvement in patients. Motor abilities is one of the domains assessed by the CGI-I scale. The CGI-I is rated on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse) as follows: 1=Very much improved; 2=Much improved; 3=Minimally improved; 4=No change; 5=Minimally worse; 6=Much worse; 7=Very much worse, where higher score indicates worse outcome. The CGI-I assessment of motor abilities was conducted by the Investigator. The number of participants in each of the 7 categories of the CGI-I for each visit is reported.
Time Frame: Months 6, 12, 18, 24, 30, 36, Last On-Treatment Visit (Up to Month 49)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Any ZX008 Open Label Dose
Number analyzed (Participants) | 399
Participants
  Month 6: Very much improved: number analyzed (Participants) | 365
  Month 6: Very much improved | 10
  Month 6: Much improved: number analyzed (Participants) | 365
  Month 6: Much improved | 33
  Month 6: Minimally improved: number analyzed (Participants) | 365
  Month 6: Minimally improved | 81
  Month 6: No change: number analyzed (Participants) | 365
  Month 6: No change | 221
  Month 6: Minimally worse: number analyzed (Participants) | 365
  Month 6: Minimally worse | 17
  Month 6: Much worse: number analyzed (Participants) | 365
  Month 6: Much worse | 1
  Month 6: Very much worse: number analyzed (Participants) | 365
  Month 6: Very much worse | 2
  Month 12: Very much improved: number analyzed (Participants) | 265
  Month 12: Very much improved | 13
  Month 12: Much improved: number analyzed (Participants) | 265
  Month 12: Much improved | 29
  Month 12: Minimally improved: number analyzed (Participants) | 265
  Month 12: Minimally improved | 52
  Month 12: No change: number analyzed (Participants) | 265
  Month 12: No change | 159
  Month 12: Minimally worse: number analyzed (Participants) | 265
  Month 12: Minimally worse | 10
  Month 12: Much worse: number analyzed (Participants) | 265
  Month 12: Much worse | 0
  Month 12: Very much worse: number analyzed (Participants) | 265
  Month 12: Very much worse | 2
  Month 18: Very much improved: number analyzed (Participants) | 226
  Month 18: Very much improved | 9
  Month 18: Much improved: number analyzed (Participants) | 226
  Month 18: Much improved | 19
  Month 18: Minimally improved: number analyzed (Participants) | 226
  Month 18: Minimally improved | 42
  Month 18: No change: number analyzed (Participants) | 226
  Month 18: No change | 133
  Month 18: Minimally worse: number analyzed (Participants) | 226
  Month 18: Minimally worse | 21
  Month 18: Much worse: number analyzed (Participants) | 226
  Month 18: Much worse | 2
  Month 18: Very much worse: number analyzed (Participants) | 226
  Month 18: Very much worse | 0
  Month 24: Very much improved: number analyzed (Participants) | 189
  Month 24: Very much improved | 7
  Month 24: Much improved: number analyzed (Participants) | 189
  Month 24: Much improved | 24
  Month 24: Minimally improved: number analyzed (Participants) | 189
  Month 24: Minimally improved | 43
  Month 24: No change: number analyzed (Participants) | 189
  Month 24: No change | 99
  Month 24: Minimally worse: number analyzed (Participants) | 189
  Month 24: Minimally worse | 13
  Month 24: Much worse: number analyzed (Participants) | 189
  Month 24: Much worse | 3
  Month 24: Very much worse: number analyzed (Participants) | 189
  Month 24: Very much worse | 0
  Month 30: Very much improved: number analyzed (Participants) | 149
  Month 30: Very much improved | 4
  Month 30: Much improved: number analyzed (Participants) | 149
  Month 30: Much improved | 19
  Month 30: Minimally improved: number analyzed (Participants) | 149
  Month 30: Minimally improved | 29
  Month 30: No change: number analyzed (Participants) | 149
  Month 30: No change | 86
  Month 30: Minimally worse: number analyzed (Participants) | 149
  Month 30: Minimally worse | 9
  Month 30: Much worse: number analyzed (Participants) | 149
  Month 30: Much worse | 1
  Month 30: Very much worse: number analyzed (Participants) | 149
  Month 30: Very much worse | 1
  Month 36: Very much improved: number analyzed (Participants) | 124
  Month 36: Very much improved | 2
  Month 36: Much improved: number analyzed (Participants) | 124
  Month 36: Much improved | 9
  Month 36: Minimally improved: number analyzed (Participants) | 124
  Month 36: Minimally improved | 27
  Month 36: No change: number analyzed (Participants) | 124
  Month 36: No change | 74
  Month 36: Minimally worse: number analyzed (Participants) | 124
  Month 36: Minimally worse | 8
  Month 36: Much worse: number analyzed (Participants) | 124
  Month 36: Much worse | 4
  Month 36: Very much worse: number analyzed (Participants) | 124
  Month 36: Very much worse | 0
  Last On-Treatment Visit: Very much improved | 12
  Last On-Treatment Visit: Much improved | 39
  Last On-Treatment Visit: Minimally improved | 89
  Last On-Treatment Visit: No change | 238
  Last On-Treatment Visit: Minimally worse | 16
  Last On-Treatment Visit: Much worse | 4
  Last On-Treatment Visit: Very much worse | 1

10. Secondary Outcome: Number of Participants With Improvement in Seizure Burden as Assessed by the Investigator
Description: The change in seizure burden from the previous visit was assessed by the investigator using following categories: <25%, ≥25%, ≥50%, ≥75%, 100% (i.e., seizure-free) improvement. Improvement in seizure burden at Baseline was based on comparison with the participant's last visit in the feeder studies (ZX008-1601, ZX008-1503, and ZX008-1602). Number of participants in each of the 5 categories is reported for each visit as compared to last visit.
Time Frame: Baseline (Day 1), Months 6, 12, 18, 24, 30, 36, Last On-Treatment Visit (Up to Month 49)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Any ZX008 Open Label Dose
Number analyzed (Participants) | 410
Participants
  Baseline: <25%: number analyzed (Participants) | 398
  Baseline: <25% | 242
  Baseline: >=25%: number analyzed (Participants) | 398
  Baseline: >=25% | 67
  Baseline: >=50%: number analyzed (Participants) | 398
  Baseline: >=50% | 42
  Baseline: >=75%: number analyzed (Participants) | 398
  Baseline: >=75% | 35
  Baseline: 100%: number analyzed (Participants) | 398
  Baseline: 100% | 12
  Month 6: <25%: number analyzed (Participants) | 381
  Month 6: <25% | 262
  Month 6: >=25%: number analyzed (Participants) | 381
  Month 6: >=25% | 51
  Month 6: >=50%: number analyzed (Participants) | 381
  Month 6: >=50% | 39
  Month 6: >=75%: number analyzed (Participants) | 381
  Month 6: >=75% | 21
  Month 6: 100%: number analyzed (Participants) | 381
  Month 6: 100% | 8
  Month 12: <25%: number analyzed (Participants) | 272
  Month 12: <25% | 191
  Month 12: >=25%: number analyzed (Participants) | 272
  Month 12: >=25% | 33
  Month 12: >=50%: number analyzed (Participants) | 272
  Month 12: >=50% | 31
  Month 12: >=75%: number analyzed (Participants) | 272
  Month 12: >=75% | 11
  Month 12: 100%: number analyzed (Participants) | 272
  Month 12: 100% | 6
  Month 18: <25%: number analyzed (Participants) | 232
  Month 18: <25% | 175
  Month 18: >=25%: number analyzed (Participants) | 232
  Month 18: >=25% | 22
  Month 18: >=50%: number analyzed (Participants) | 232
  Month 18: >=50% | 26
  Month 18: >=75%: number analyzed (Participants) | 232
  Month 18: >=75% | 3
  Month 18: 100%: number analyzed (Participants) | 232
  Month 18: 100% | 6
  Month 24: <25%: number analyzed (Participants) | 193
  Month 24: <25% | 144
  Month 24: >=25%: number analyzed (Participants) | 193
  Month 24: >=25% | 24
  Month 24: >=50%: number analyzed (Participants) | 193
  Month 24: >=50% | 15
  Month 24: >=75%: number analyzed (Participants) | 193
  Month 24: >=75% | 6
  Month 24: 100%: number analyzed (Participants) | 193
  Month 24: 100% | 4
  Month 30: <25%: number analyzed (Participants) | 148
  Month 30: <25% | 115
  Month 30: >=25%: number analyzed (Participants) | 148
  Month 30: >=25% | 14
  Month 30: >=50%: number analyzed (Participants) | 148
  Month 30: >=50% | 11
  Month 30: >=75%: number analyzed (Participants) | 148
  Month 30: >=75% | 7
  Month 30: 100%: number analyzed (Participants) | 148
  Month 30: 100% | 1
  Month 36: <25%: number analyzed (Participants) | 128
  Month 36: <25% | 99
  Month 36: >=25%: number analyzed (Participants) | 128
  Month 36: >=25% | 13
  Month 36: >=50%: number analyzed (Participants) | 128
  Month 36: >=50% | 9
  Month 36: >=75%: number analyzed (Participants) | 128
  Month 36: >=75% | 6
  Month 36: 100%: number analyzed (Participants) | 128
  Month 36: 100% | 1
  Last On-Treatment Visit: <25% | 315
  Last On-Treatment Visit: >=25% | 41
  Last On-Treatment Visit: >=50% | 29
  Last On-Treatment Visit: >=75% | 17
  Last On-Treatment Visit: 100% | 8

ADVERSE EVENTS:
Time Frame: From First dose of ZX008 (in study EP0215 [ZX008-1900]) to Cardiac Follow-up after ZX008 treatment (Up to 6 Years, 17 Days)
Description: TEAEs were defined as AE that began on or after the first day of treatment with ZX008 in Study EP0215 (ZX008-1900) (NCT03936777) or that occurred prior to first ZX008 treatment in Study EP0215 (ZX008-1900) but increased in severity after treatment in Study EP0215 (ZX008-1900) began. Events recorded at Follow-up/Cardiac Follow-up were considered treatment emergent. Safety analysis set consisted of participants who received at least one dose of ZX008 during the open label extension.
Arm/Group | Any ZX008 Open Label Dose
All-Cause Mortality (participants affected / at risk) | 3/412
Serious Adverse Events (participants affected / at risk) | 67/412
Other Adverse Events (participants affected / at risk) | 204/412
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Any ZX008 Open Label Dose (N=412)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (3)
Cardiac arrest (Cardiac disorders) | 1 (1)
Non-compaction cardiomyopathy (Congenital, familial and genetic disorders) | 1 (1)
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 2 (2)
Complication associated with device (General disorders) | 1 (2)
Gait disturbance (General disorders) | 1 (1)
Gait inability (General disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Pneumonia (Infections and infestations) | 8 (8)
Appendicitis (Infections and infestations) | 2 (2)
Corona virus infection (Infections and infestations) | 2 (2)
Pneumonia viral (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 1 (2)
Cellulitis of male external genital organ (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Dengue haemorrhagic fever (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Legionella infection (Infections and infestations) | 1 (1)
Nasal abscess (Infections and infestations) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1)
Craniofacial fracture (Injury, poisoning and procedural complications) | 1 (1)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Spinal column injury (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Traumatic renal injury (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 1 (1)
Seizure (Nervous system disorders) | 17 (22)
Status epilepticus (Nervous system disorders) | 9 (10)
Seizure cluster (Nervous system disorders) | 2 (2)
Epilepsy (Nervous system disorders) | 1 (4)
Altered state of consciousness (Nervous system disorders) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Parkinsonism (Nervous system disorders) | 1 (1)
Petit mal epilepsy (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Thalamus haemorrhage (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Aggression (Psychiatric disorders) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1)
Intentional self-injury (Psychiatric disorders) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 5 (11)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Any ZX008 Open Label Dose (N=412)
Diarrhoea (Gastrointestinal disorders) | 29 (36)
Pyrexia (General disorders) | 53 (86)
Corona virus infection (Infections and infestations) | 84 (99)
Nasopharyngitis (Infections and infestations) | 49 (69)
Upper respiratory tract infection (Infections and infestations) | 23 (28)
Decreased appetite (Metabolism and nutrition disorders) | 25 (30)
Seizure (Nervous system disorders) | 52 (69)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-09-22): https://cdn.clinicaltrials.gov/large-docs/77/NCT03936777/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-27): https://cdn.clinicaltrials.gov/large-docs/77/NCT03936777/SAP_001.pdf